CLINICAL TRIAL: NCT05454267
Title: Early Detection of Vaping-related Vascular Diseases
Acronym: ENDS
Status: Recruiting | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: Florida Department of Health (Other Government)
Responsible Party: Principal Investigator, Adam Wanner, Professor of Medicine, University of Miami
Other Study IDs: 20211060
Record Dates: First submitted 2022-06-30; First posted 2022-07-12 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Vaping; Blood Vessel Injury
MeSH Terms: conditions — Vaping; Vascular System Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Oral swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Healthy Volunteer Group: Participants who have never smoked or vaped
- High Frequency Vaping Group: Participants who vape >20 days per month.
- Low-Frequency Vaping Group: Participants who vape < 20 days per month

SUMMARY:
The purpose of this study is to determine how vaping affects blood vessels, in particular if early damage occurs in the lung vessels.

ELIGIBILITY:
Inclusion Criteria:

Vapers Group:

1. Current electronic cigarette (EC) Puff Bar users defined as using EC either daily or occasionally in the past 30 days for at least 6 months, and with 5% nicotine concentration pods.
2. Adults aged 18-40 years

Healthy Group:

1. Healthy never smokers, never vapers
2. Adults aged 18-40 years

Exclusion Criteria:

1. Current or past smoking of tobacco cigarette (TC) or other tobacco/nicotine products (e.g., smokeless tobacco, Hookah) or marijuana will be excluded from the study.
2. Subjects with self-reported history of chronic health problems including asthma, chronic obstructive pulmonary disease (COPD), morbid obesity (BMI>40 kg/m2), hypertension or diabetes
3. Pregnant or breastfeeding women

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy non smokers and vapers residing in Florida
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Airway blood flow reactivity (QAW) | Up to 1 week
  QAW will be measured via soluble gas uptake method
Pulmonary vascular resistance (PVR) | Up to 4 weeks
  PVR will be measured via echocardiography
Flow-mediated vasodilation (FMD) | Up to 4 weeks
  FMD will be measured by blood pressure cuff deflation using ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Adam Wanner, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Health System, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No